CLINICAL TRIAL: NCT06862167
Title: Comparative Study Between Desarda's Technique Versus Lichtenstein's Technique Hernia Repair in Management of Elective Non-complicated Inguinal Hernia (Randomized Controlled Trial)
Brief Title: Desarda's Technique Versus Lichtenstein's Technique Hernia Repair in Management of Elective Non-Complicated Inguinal Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Salah, Lecturer in General Surgery Department, Minia University, Minia, Egypt, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1240/08/2024
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Desarda's Technique; Lichtenstein's Technique; Hernia Repair; Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desarda's technique group (Experimental): Patients will undergo Desarda's technique.
  Interventions: Procedure: Desarda's technique
- Lichtenstein's technique group (Active Comparator): Patients will undergo Lichtenstein's technique.
  Interventions: Procedure: Lichtenstein's technique

INTERVENTIONS:
Procedure: Desarda's technique — Patients will undergo Desarda's technique.
  Arms: Desarda's technique group
Procedure: Lichtenstein's technique — Patients will undergo Lichtenstein's technique.
  Arms: Lichtenstein's technique group

SUMMARY:
This study aims to compare Desarda's technique and Lichtenstein's technique of hernia repair in managing elective, non-complicated inguinal hernia.

DETAILED DESCRIPTION:
Mesh prosthesis was introduced to hernial surgery as a magic solution for any inguinal hernia, and it has significant advantages (Simplicity of the procedure, Mesh is cheap, and has a low recurrence rate). Still, mesh induces fibrosis that can lead to stiffness and foreign body sensation, which become a source of agony for the patient. Mesh infection is one of the serious complications that can lead to the removal of the mesh and long-term terms morbidity from Lichtenstein hernia repairs, such as Vas entrapment and Chronic groin pain.

Desarda technique requires no extensive dissection or only suturing; no mesh is needed, and it is easy to learn. It is still ferrated and determined the optimum procedure to treat an inguinal hernia. It is a straightforward operation that avoids the risks of mesh implantation, has a low recurrence rate, and can be done by non-consultant staff.

ELIGIBILITY:
Inclusion Criteria:

* Above 14 years of age.
* With reducible non-complicated inguinal or inguinoscrotal hernia; unilateral or bilateral

Exclusion Criteria:

* Obstructive uropathy or chronic obstructive pulmonary disease because they are contraindications to elective hernia surgery. They are associated with definite poor outcomes, such as high recurrence rates.
* Unfit patients for surgery
* Patients with strangulated hernia.
* Recurrent Hernias.
* Per operative finding of separated, thin, and/or weak external oblique aponeurosis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | 1 year postoperatively
  Incidence of postoperative complications such as groin pain, hemorrhage, orchitis, testicular atrophy, and seroma will be recorded.

SECONDARY OUTCOMES:
Time till stop of postoperative analgesic | 30 days postoperatively
  Stop of postoperative analgesic (Within 3 days, 3 to 6 days, More than 6 days)
Return to normal activity | 30 days postoperatively
  Return to normal activity will be recorded from 1 to 7 days, 8 to 15 days, and 16 to 30 days postoperatively.
Incidence of recurrence | 1 year postoperatively
  Incidence of recurrence will be recorded within 1 year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.